CLINICAL TRIAL: NCT02078557
Title: A Multiple Dose Titration Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8892 in Patients With Pulmonary Hypertension and Left Heart Disease
Brief Title: A Multiple Dose Titration Study of MK-8892 in Participants With Pulmonary Hypertension and Left Heart Disease (MK-8892-007)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8892-007; 2013-004639-55 (EudraCT Number); MK-8892-007 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Hypertension; Left Heart Disease
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-8892 (Experimental): Starting dose of 1 mg daily (oral); the dose may be titrated up on the 8th, 15th, and 22nd day of treatment to 2 mg, 3 mg, or 4 mg, respectively, for the duration of the study (28 days) as tolerated. For participants who reach one or more of the down-dosing criteria, there is an opportunity to decrease the dose back to a previously well-tolerated dose level, or to ½ of the starting dose.
  Interventions: Drug: MK-8892

INTERVENTIONS:
Drug: MK-8892

SUMMARY:
This study will assess multiple doses of MK-8892 administered to participants with pulmonary hypertension "out of proportion" (PHOOP) and heart failure with reduced left ventricular ejection fraction (rEF). It is hypothesized that generally safe and well tolerated multiple doses of MK-8892 will achieve a true reduction from baseline in pulmonary vascular resistance (PVR) greater than 12%.

Sixteen participants with PHOOP/rEF were to receive multiple doses of MK-8892 titrated to the highest tolerated dose for each participant (up to 4 mg daily), and to undergo evaluation for safety and systemic hemodynamics and cardiac function. Only 4 participants were enrolled and completed the study due to a strategic business decision by the sponsor to terminate the clinical conduct of all MK-8892 ongoing trials including this trial.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension (out of proportion, PHOOP) and heart failure with reduced left ventricular ejection fraction (PHOOP/rEF)
* If female, cannot be pregnant or breastfeeding. Females of reproductive potential must agree to agree to use (and/or have their partner use) two (2) acceptable methods of birth control throughout the study and until 2 weeks after the last dose of study drug is administered
* Body mass index (BMI) <=35 kg/m^2 and and <=18 kg/m^2
* Has World Health Organization (WHO) Group 2 pulmonary hypertension (PAH)
* Stable heart failure on optimal medical therapy with no hospitalizations for congestion due to heart failure within the previous 3 months

Exclusion Criteria:

* Primary pulmonary arterial hypertension or veno-occlusive disease (WHO Group 1), or pulmonary hypertension secondary to other causes (WHO Groups 3 -5) including but not limited to autoimmune disease, connective tissue disease, and Eisenmenger syndrome
* Currently treatment with or anticipates use of nitrate, phosphodiesterase type 5 (PDE5) inhibitor, or medications known to induce or inhibit cytochrome P450 3A4 (CYP3A4) metabolism, and cannot be transitioned off of this therapy for >=7 days prior to dosing and through completion of this study
* Symptoms of coronary artery disease requiring therapy with nitrates, within the past 3 months
* Severe aortic or mitral stenosis, or severe aortic, mitral, or tricuspid insufficiency.
* Significant carotid artery disease
* Restrictive, infiltrative (e.g., amyloidosis) or hypertrophic cardiomyopathy
* Mentally or legally institutionalized or incapacitated, has significant emotional problems at the time of pre study (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years. Subjects who have had situational depression may be enrolled in the study at the discretion of the investigator.
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine (not including diabetes mellitus), gastrointestinal, hematological, hepatic (not including chronic Hepatitis C), immunological (not including chronic human immunodeficiency virus [HIV]), respiratory, or genitourinary abnormalities or diseases. Participants with a history of childhood asthma may be enrolled in the study at the discretion of the investigator. Participants with controlled hypertension are allowed to be enrolled.
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the dose of study drug, throughout the study (including washout intervals between treatment periods), until the post study visit. There may be certain medications that will be permitted.
* Consumes excessive amounts of alcohol, defined as greater than 5 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Major surgery or donated blood within 8 weeks prior to the pre study (screening) visit
* Participated in another investigational study within 4 weeks prior to the pre study (screening) visit
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Uses illicit drugs or has a history of drug (including alcohol) abuse within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2014-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8892: MK-8892 once daily for 28 days titrated to the highest tolerated dose per participant (up to 4 mg).
Period: Overall Study
Arm/Group | MK-8892
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-8892
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Pulmonary Vascular Resistance (PVR)
Description: Pulmonary vascular resistance (PVR) is the general pressure which the right ventricle must counteract to pump blood through the lungs. PVR was measured by right heart catheterization performed prior to dosing at baseline (Day 1) and 4 hours postdose on Day 28. Percentage change in PVR from baseline at Day 28 was calculated as [(Baseline-Day 28)/Baseline]. Standard deviation is reported as a percentage.
Time Frame: Baseline and Day 28
Population: The population for the efficacy analysis consisted of all participants who completed the 28 days of study.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | MK-8892
Number analyzed (Participants) | 4
Percentage change | -51 (199)

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or disease temporally associated with the use of the study drug or a study procedure, whether or not considered related to the study drug or study procedure. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse event.
Time Frame: Up to 42 days
Population: All participants who received at least one dose of the investigational drug
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8892
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 28 days
Population: All participants who received at least one dose of the investigational drug
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8892
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: All participants who received at least one dose of the investigational drug
Arm/Group | MK-8892
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.